CLINICAL TRIAL: NCT06778083
Title: STI Prophylaxis and Emergence of Antimicrobial Resistance
Acronym: SPEAR
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 174194; REC Ref: 24/EM/0282 (Other: NHS Health Research Authority)
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Sexually Transmitted Infection (STI) Prevention; Antibiotic Prophylaxis; Antibiotic Resistance, Bacterial; Microbiome; Doxycycline
Keywords: DoxyPEP; STI Prophylaxis; Doxycycline; STI Prevention; Antimicrobial Resistance; Antibiotic Resistance; Microbiome; Men-who-have-sex-with-men
MeSH Terms: conditions — Sexually Transmitted Diseases; Homosexuality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Oropharyngeal Swab
  2. Stool Sample
  Samples will undergo bacterial DNA extraction and host cell depletion, following by metagenomic sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DoxyPEP users: Previous use of doxycycline post-exposure prophylaxis within 3 months of baseline visit.
- Doxycycline treatment: Previous use of doxycycline for STI treatment within 3 months of baseline visit.
  Once enrolled all participants may use doxycycline post-exposure prophylaxis.
- No antibiotics: No antibiotics within previous 3 months of baseline visit. Once enrolled all participants may use doxycycline post-exposure prophylaxis.

SUMMARY:
The goal of this observational study is to understand the risk of antibiotic resistance and changes in the human microbiome (bacteria that live inside and on us), if people use antibiotics to prevent sexually transmitted infections (STI prophylaxis, doxycycline post-exposure prophylaxis, or 'doxyPEP'). The study will assess how easy and acceptable it is to find antibiotic resistance and microbiome changes in the throats and guts of men-who-have-sex-with-men (MSM) who use STI prophylaxis.

The study will recruit 108 MSM who are using and not using STI prophylaxis. Participants will visit the clinic every 6 months. At each visit, they will provide a throat swab and stool sample, and complete a questionnaire. DNA of the bacteria from the samples will be analysed to identify the bacteria and look for antibiotic resistance.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years.
* Identifies as a man (cis or trans).
* Has sex with men.
* Able to provide informed consent.

Exclusion Criteria:

* Use of an antibiotic other than doxycycline in the 3 months prior to enrolment
* Currently being treated for an STI with doxycycline
* Use of doxycycline within the prior 3 months for an indication other than STI treatment or STI prevention.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men-who-have-sex-with-men
Study Population: Men-who-have-sex-with men aged ≥ 18 years living in the United Kingdom. Target of 108 participants, with minimum 40 participants living with HIV.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Detection of antimicrobial resistance genes of interest and characterisation of microbiome | From enrolment to 12 months
  The successful detection of antimicrobial resistance genes of interest (tetracycline and other antibiotic classes) and identification of bacterial species (microbiome) and in the oropharynx and gastrointestinal tract.

SECONDARY OUTCOMES:
Detection of differences in prevalence of antimicrobial resistance genes of interest between people using and not using antibiotic STI prophylaxis. | From enrolment to 12 months
Detection of differences in microbiome between people using and not using antibiotic STI prophylaxis. | From enrolment to 12 months
Change over time in prevalence of antimicrobial resistance genes of interest between people using and not using antibiotic STI prophylaxis. | From enrolment to 12 months
Change over time in microbiome between people using and not using antibiotic STI prophylaxis. | From enrolment to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Central and North West London NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kohli M, Reid D, Pulford CV, Howarth A, Brown J, Mohammed H, Hughes G, Mercer CH, Saunders J. Choice of antibiotics for prophylaxis of bacterial STIs among individuals currently self-sourcing. Sex Transm Infect. 2022 Mar;98(2):158. doi: 10.1136/sextrans-2021-055310. Epub 2021 Dec 6. No abstract available. PMID 34873029
- [Background] Kohli M, Medland N, Fifer H, Saunders J. BASHH updated position statement on doxycycline as prophylaxis for sexually transmitted infections. Sex Transm Infect. 2022 May;98(3):235-236. doi: 10.1136/sextrans-2022-055425. No abstract available. PMID 35414633
- [Background] Chu VT, Glascock A, Donnell D, Grabow C, Brown CE, Ward R, Love C, Kalantar KL, Cohen SE, Cannon C, Woodworth MH, Kelley CF, Celum C, Luetkemeyer AF, Langelier CR. Impact of doxycycline post-exposure prophylaxis for sexually transmitted infections on the gut microbiome and antimicrobial resistome. Nat Med. 2025 Jan;31(1):207-217. doi: 10.1038/s41591-024-03274-2. Epub 2024 Oct 3. PMID 39363100
- [Background] Molina JM, Charreau I, Chidiac C, Pialoux G, Cua E, Delaugerre C, Capitant C, Rojas-Castro D, Fonsart J, Bercot B, Bebear C, Cotte L, Robineau O, Raffi F, Charbonneau P, Aslan A, Chas J, Niedbalski L, Spire B, Sagaon-Teyssier L, Carette D, Mestre SL, Dore V, Meyer L; ANRS IPERGAY Study Group. Post-exposure prophylaxis with doxycycline to prevent sexually transmitted infections in men who have sex with men: an open-label randomised substudy of the ANRS IPERGAY trial. Lancet Infect Dis. 2018 Mar;18(3):308-317. doi: 10.1016/S1473-3099(17)30725-9. Epub 2017 Dec 8. PMID 29229440
- [Background] Molina JM, Bercot B, Assoumou L, Rubenstein E, Algarte-Genin M, Pialoux G, Katlama C, Surgers L, Bebear C, Dupin N, Ouattara M, Slama L, Pavie J, Duvivier C, Loze B, Goldwirt L, Gibowski S, Ollivier M, Ghosn J, Costagliola D; ANRS 174 DOXYVAC Study Group. Doxycycline prophylaxis and meningococcal group B vaccine to prevent bacterial sexually transmitted infections in France (ANRS 174 DOXYVAC): a multicentre, open-label, randomised trial with a 2 x 2 factorial design. Lancet Infect Dis. 2024 Oct;24(10):1093-1104. doi: 10.1016/S1473-3099(24)00236-6. Epub 2024 May 23. PMID 38797183
- [Background] Luetkemeyer AF, Donnell D, Dombrowski JC, Cohen S, Grabow C, Brown CE, Malinski C, Perkins R, Nasser M, Lopez C, Vittinghoff E, Buchbinder SP, Scott H, Charlebois ED, Havlir DV, Soge OO, Celum C; DoxyPEP Study Team. Postexposure Doxycycline to Prevent Bacterial Sexually Transmitted Infections. N Engl J Med. 2023 Apr 6;388(14):1296-1306. doi: 10.1056/NEJMoa2211934. PMID 37018493

DOCUMENTS (1):
  • Study Protocol (2024-12-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT06778083/Prot_000.pdf